CLINICAL TRIAL: NCT00188071
Title: Postoperative Pain After Medical Abortion Under Local Anesthesia : a Prospective and Randomized Trial Comparing Several Analgesic Regimen
Brief Title: Postoperative Pain After Medical Abortion Under Local Anesthesia : Comparison of Several Analgesic Regimen
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Angers (Other Government)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CP 02-02
Record Dates: First submitted 2005-09-12; First posted 2005-09-16 (Estimated); Last update posted 2017-11-01 (Actual); Status verified 2005-09

CONDITIONS: Abortion, Induced
Keywords: medical abortion; analgesia
MeSH Terms: conditions — Agnosia | interventions — Acetaminophen; Ketoprofen

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Drug: paracetamol
Drug: ketoprofen
Drug: ketoprofen + paracetamol

SUMMARY:
* To compare postoperative analgesia by paracetamol 1gr or ketoprofen 100 mg or the combination of these two analgesics
* each treatment beeing allocated by randomization

DETAILED DESCRIPTION:
* 240 pregnant women who undewent a medical abortion by aspiration, under local anesthesia, (day case surgery) were enrolled after informed consent and signed approval
* according to randomization, they received one hour before medical abortion procedure performed under local anesthesia of the cervix, one of these three diffrente analgesics :

  * paracetamol 1 gr
  * ketoprofen 100 mg
  * the association of both Postprocedure pain was recorded, by nurse, using a visual analog scale (VAS), 7 times before and after the procedure, until the discharge of the patient.
* if VAS was above 40 on two consecutive measurements a morphine injection was given.
* the number and total amount of morphine was recorded.
* satisfaction was recorded within the 3 postoperative day by a telephone inquiry.

ELIGIBILITY:
Inclusion Criteria:

* pregnant women
* medical abortion performed in day case surgery under local anesthesia
* informed written consent

Exclusion Criteria:

* under 18 year old

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 240
Dates: Start 2002-09; Study Completion 2003-08

PRIMARY OUTCOMES:
postoperative pain rating

SECONDARY OUTCOMES:
morphine consumption
patient satisfaction

CONTACTS AND LOCATIONS:
Overall Officials: Jean Claude Granry, MD, Study Chair — University hospital, Angers, FRANCE; Emmanuel Mucci, MD, Principal Investigator — University hospital, Angers, FRANCE; Christine Monrigal, MD, Study Director — Dept of Anesthesia, CHU, Angers - France
Locations (1):
- Dept of Anesthesia - CHU, Angers, France